CLINICAL TRIAL: NCT02363621
Title: Evaluation of Inflammation and Pain Post Injection of Ranibizumab vs. Aflibercept in Patients With Diabetic Macular Edema
Brief Title: Evaluation of Inflammation and Pain Post Injection of Ranibizumab vs Aflibercept in Patients With DME
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arshad Khanani (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Arshad Khanani, Vitreo-Retinal Diseases and Surgery, Sierra Eye Associates
Organization: Sierra Eye Associates (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ML29634
Record Dates: First submitted 2015-02-02; First posted 2015-02-16 (Estimated); Results first posted 2019-04-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Ranibizumab; aflibercept

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Ranibizumab 0.3 Intravitreal injection (Active Comparator): Intravitreal injection of Ranibizumab 0.3 mg once
  Interventions: Drug: Ranibizumab 0.3 mg
- Aflibercept 2.0 mg intravitreal injection (Active Comparator): Intravitreal Aflibercept 2.0 mg once
  Interventions: Drug: Aflibercept 2.0 mg

INTERVENTIONS:
Drug: Ranibizumab 0.3 mg — Ranibizumab 0.3 mg Patient will receive intravitreal injection of Ranibizumab 0.3 mg
  Other Names: Lucentis
  Arms: Ranibizumab 0.3 Intravitreal injection
Drug: Aflibercept 2.0 mg — Patient will receive intravitreal injection of Aflibercept 2.0 mg
  Other Names: Eylea
  Arms: Aflibercept 2.0 mg intravitreal injection

SUMMARY:
This study is designed to compare the post injection inflammation and pain seen after intravitreal injections of ranibizumab 0.3mg and aflibercept 2.0mg in patients with DME.

The investigators will be evaluating patients (1-7 days) post injections for:

1. Intraocular inflammation (defined as anterior chamber and/or vitreous cells 2. Pain (as measured on a standardized pain scale).

DETAILED DESCRIPTION:
This is an open-label, Phase II study of post injection pain and inflammation after intravitreally administered ranibizumab and aflibercept in 100 subjects with Diabetic Macular Edema. Treatment naïve and experienced patients will be enrolled. Treatment experienced patients with history of anti-vegf injections will be eligible as long as they have not received any intravitreal injection in the 3 months prior to the study visit. Patients will be randomized to receive either Lucentis 0.3 mg or Eylea 2.0 mg, and followed for a week. A non-injecting masked physician who is blinded to the treatment drug will evaluate the patient at baseline before the injection and then within 1-2 days and 5-7 days after the injection for anterior chamber and vitreous cells using slit lamp examination and indirect ophthalmoscopy. Pain will also be recorded at these visits using a standardized pain scale.

Consented, enrolled subjects will receive open-label intravitreal injection of either 0.3 mg ranibizumab or 2.0 mg aflibercept. A standard intravitreal injection protocol will be followed. Patients will be revaluated at baseline, 1-2 days and 5-7 days post injections. A non-injecting physician will evaluate the patients for anterior chamber and vitreous inflammation; this physician will be blinded about the specific treatment. Anterior chamber inflammation is described as any cell or flare in the anterior chamber. These will be evaluated using Standardization of Uveitis Nomenculature (SUN) working group classifications. Pain score will be evaluated using a Numerical Rating Scale.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be eligible if the following criteria are met:
* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 21 years
* Exam and OCT confirming Diabetic Macular Edema
* Visual Acuity of 20/400 or better
* No history of post injection pain or inflammation in the past

Exclusion Criteria:

* Subjects who meet any of the following criteria will be excluded from this study
* History of Endophthalmitis in either eye
* Current inflammation in either eye
* Uncontrolled or symptomatic Dry Eye Syndrome
* Intravitreal injection less than 3 months ago
* History of Anterior or Posterior Uveitis
* History of post injection pain with prior treatments
* Recent thromboembolic event (<3 months)
* Pregnancy (positive pregnancy test) or lactation
* Premenopausal women not using adequate contraception.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2015-01; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arshad Khanani, MD, Principal Investigator — Sierra Eye Associates
Locations (1):
- Sierra Eye Associates, Reno, Nevada, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ranibizumab 0.3 Intravitreal Injection | Aflibercept 2.0 mg Intravitreal Injection
Started | 51 | 50
Completed | 50 | 50
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: Patients with diabetic macular edema
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranibizumab 0.3 Intravitreal Injection | Aflibercept 2.0 mg Intravitreal Injection | Total
Number analyzed (Participants) | 51 | 50 | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 26 | 55
  >=65 years | 22 | 24 | 46
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 21 | 39
  Male | 33 | 29 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 12 | 26
  Not Hispanic or Latino | 37 | 38 | 75
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 4 | 1 | 5
  Black or African American | 2 | 2 | 4
  White | 40 | 44 | 84
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 51 | 50 | 101
Diabetic Macular Edema [Count of Participants; unit: Participants] — Diabetic Macular edema as seen on OCT and exam.
  Participants | 51 | 50 | 101

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Intraocular Inflammation
Description: Number of participants with intraocular inflammation as seen on slide lamp and dilated fundus exam.
Time Frame: 24 to 48 hours (visit #1)
Measure: Count of Participants; unit: Participants
Arm/Group | Ranibizumab 0.3 Intravitreal Injection | Aflibercept 2.0 mg Intravitreal Injection
Number analyzed (Participants) | 50 | 50
Participants | 6 | 10

2. Primary Outcome: Number of Participants With Intraocular Inflammation
Description: Number of Participants With Intraocular Inflammation as seen on slit lamp and dilated fundus exam
Time Frame: 5 to 7 days (visit #2)
Population: Inflammation 5 to 7 days after injection
Measure: Count of Participants; unit: Participants
Arm/Group | Ranibizumab 0.3 Intravitreal Injection | Aflibercept 2.0 mg Intravitreal Injection
Number analyzed (Participants) | 50 | 50
Participants | 1 | 3

3. Secondary Outcome: Number of Participants With Post Injection Pain Above 0 on a 11 Point Pain Scale.
Description: Pain score rated on a 11 point numerical rating from 0-10 administered to each patient verbally at visit #1 and visit #2.
  0 = no pain 10 = severe pain
Time Frame: 24 to 48 hours visit #1 and 5 to 7 days visit #2
Measure: Count of Participants; unit: Participants
Arm/Group | Ranibizumab 0.3 Intravitreal Injection | Aflibercept 2.0 mg Intravitreal Injection
Number analyzed (Participants) | 50 | 50
Participants
  24 to 48 hours visit #1 | 28 | 28
  5 to 7 days visit #2 | 10 | 5

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Ranibizumab 0.3 Intravitreal Injection | Aflibercept 2.0 mg Intravitreal Injection
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/50
Other Adverse Events (participants affected / at risk) | 6/51 | 10/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranibizumab 0.3 Intravitreal Injection (N=51) | Aflibercept 2.0 mg Intravitreal Injection (N=50)
anterior chamber inflammation (Eye disorders) | 6 (6) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-12-14): https://cdn.clinicaltrials.gov/large-docs/21/NCT02363621/Prot_SAP_000.pdf